CLINICAL TRIAL: NCT04709913
Title: A Double-blind, Sponsor-Open, Placebo-controlled, Phase I Study of the Safety, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of HU6 in High BMI Volunteers
Brief Title: Multiple Ascending Dose Study of HU6 in High BMI Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-HU6-102
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: The study will be conducted in one phase: a single dose, dose escalation phase in up to 4 cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment: HU6 Planned doses of HU6; N = 32 (Active Comparator): Drug = HU6 HU6 is designed to reduce the steatosis, inflammation, fibrosis and hepatocyte injury in Noncirrhotic Nonalcoholic Steatohepatitis (NASH)
  Interventions: Drug: HU6
- Placebo Comparator Non-active study drug N = 8 (Placebo Comparator): Placebo Comparator, non-active study drug.
  Interventions: Drug: HU6

INTERVENTIONS:
Drug: HU6 — HU6 is designed to reduce the steatosis, inflammation, fibrosis and hepatocyte injury in Noncirrhotic Nonalcoholic Steatohepatitis (NASH)

SUMMARY:
This is a 14-day multiple ascending dose trial in high BMI volunteers in up to 4 cohorts of 10 high BMI volunteers each consisting of 8 receiving HU6 and 2 receiving placebo. Upon review of the safety and PK data, it may be decided to expand the current cohort size and/or dose escalate to the next cohort. In addition, the sponsor may elect not to enroll all 4 cohorts based on safety and/or PK and/or PD data, or enlist an additional cohort at a higher dose if deemed safe.

DETAILED DESCRIPTION:
This is a 14-day multiple ascending dose trial in high BMI volunteers in up to 4 cohorts of 10 high BMI volunteers each consisting of 8 receiving HU6 and 2 receiving placebo. Upon review of the safety and PK data, it may be decided to expand the current cohort size and/or dose escalate to the next cohort. In addition, the sponsor may elect not to enroll all 4 cohorts based on safety and/or PK and/or PD data, or enlist an additional cohort at a higher dose if deemed safe.

Double-blind dosing will occur in cohorts 1 through 4. In these cohorts, 8 subjects will receive HU6 and 2 will receive matching placebo. Doses will escalate and may be modified based on results of safety and pharmacokinetic evaluation conducted after each cohort.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female between 18 and 45 years of age, inclusive, at time of informed consent.

  1. Female subjects of childbearing potential must be non-lactating, not pregnant as confirmed by a negative urine pregnancy test at Screening and admission to Clinical Research Unit, and using, and agree to continue using, an effective method of contraception for at least 4 weeks or barrier method for 2 weeks prior to first study drug administration until 30 days after the last dose of study drug.
  2. Female subjects of non-childbearing potential must be surgically sterile (e.g., hysterectomy, bilateral tubal ligation, oophorectomy) or post-menopausal (no menses for >1 year with follicle stimulating hormone >40 U/L at Screening).
  3. Female subjects of childbearing potential must not donate ova during the study and for at least 30 days after the last dose of study drug.
  4. Male subjects who have not had a vasectomy and/or subjects who have had a vasectomy but have not had 2 post surgery negative tests for sperm must agree to use an acceptable method of contraception from time of first dose of study drug until 30 days after the last dose of the study drug, and to not donate sperm during the study and for at least 30 days after the last dose of study drug.

     2. Healthy per investigator judgment as documented by medical history, physical examination, vital sign assessments, 12-lead ECG, clinical laboratory assessments, and general observations.

  <!-- -->

  1. At Screening, abnormalities or deviations outside the normal ranges for any clinical assessments that are considered clinically significant by the Investigator (laboratory tests, ECG, vital signs) may be repeated once at the discretion of the Investigator(s), and results that continue to be outside the normal ranges must be judged by the investigator to be not clinically significant and acceptable for study participation.
  2. On admission to Clinical Research Unit, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, must be within the upper limits of the normal range. Subjects with isolated elevation of bilirubin and presumptive Gilbert's syndrome are permissible. All other laboratory test results that are outside the reference range on admission to CRU and judged by the investigator to be not clinically significant may optionally be repeated. Results that continue to be outside the reference range must be judged by the investigator to be not clinically significant and acceptable for study participation.
  3. Subject must demonstrate clinical euthyroidism as assessed by a thyroid profile utilizing TSH and Free T4 testing at screening.

     3. Body mass index ≥35.0 kg/m2. 4. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

     5. Willing and able to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the investigator, which may impact safety. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening.
2. Any surgical or medical condition or history that, in the opinion of the investigator, may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to, gastric bypass surgery or significant small bowel resections.
3. Contraindication to study drug or its excipients and/or history of allergic or anaphylactic reactions.
4. Resting heart rate <45 or >110 bpm; blood pressure < 90 or >160 mm Hg systolic, or <50 or >110 diastolic.
5. Waist circumference ≤38.0 inches for men and ≤33.0 inches for women.
6. On screening ECG and by history:

   1. A marked baseline prolongation of QT/QTcF interval (e.g., repeated demonstration of a QTcF interval > 450 msec for males and >470 msec for females).
   2. A history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) or a family history of sudden cardiac death of unknown origin.
7. Taking any of the following prohibited medications:

   a. Limited background prescription medications are permitted to manage complications of obesity, but any drug known to inhibit or induce cytochrome P450 (CYP) enzymes and/or P-glycoprotein including St. John's wort (Hypericum perforatum) within 14 days or 5 half-lives (whichever is longer) prior to admission to CRU, is prohibited. Also prohibited is the use of concomitant medications that prolong the QT/QTc interval identified in the https://crediblemeds.org/ website list category of 'Known Risk'. Over the counter multi-vitamin supplements, including products with CBD, or any non-prescription products (including herbal-containing preparations) are prohibited within 14 days prior to admission to CRU or during the conduct of the trial. Acetaminophen may be taken during screening, but should not receive a dose within 24 hours of admission to the CRU.

   i) Exception: hormonal contraceptives and hormone replacement therapies (oral, injectable, transdermal or implanted) are permitted.
8. History of significant drug abuse within one year prior to Screening or frequent use of soft drugs (such as marijuana) within 3 months prior to the Screening visit, or hard drugs (such as cocaine, phencyclidine [PCP], opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
9. History of regular alcohol consumption exceeding 14 drinks/week [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months of Screening.
10. Positive urine drug or urine alcohol test at Screening or on admission to CRU.
11. Current nicotine use or vaping regularly more than 5 cigarettes or the equivalent per week. Use of nicotine patches for smoking cessation is not permitted within 7 days of dosing.
12. Consumed any food or drink/beverage containing grapefruit or grapefruit juice, apple or orange juice, pomelo juice, star fruit, Seville or Moro (blood) orange products within 6 days before admission to CRU. Vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard), food containing poppy seeds (e.g., muffins, bagels, and cakes) must not be consumed within 24 hours before admission to CRU.
13. Positive test results of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV1/2) antibody.
14. Diabetes reflected by a fasting plasma glucose level of ≥126 mg/dL and a reflex HbA1c of ≥6.5%.
15. Neutropenia, defined as absolute neutrophil count ≤1000/microL.
16. Participation in another clinical trial at the time of screening or exposure to any investigational agent, including topical, within 30 days or 5 half-lives prior to admission to CRU, whichever is longer.
17. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
18. Received a tattoo or body piercing (including ear piercings) within 2 months prior to Day 1, and/or significant open wound that may result in risk of infection.
19. Having a condition that the investigator believes would interfere with his/her ability to provide written informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk. Subjects with a history of hypo- or hyperthyroidism, peripheral neuropathy, malignant hyperthermia, cataracts or chronic recurrent rash that is considered clinically significant by the investigator are excluded.
20. Must not be claustrophobic or have a history of claustrophobia, or intolerance of closed or small spaces.
21. Familial (mother/father/sibling) and/or personal history of retinal detachment any time in the past.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Assess the dose relationship of PK Parameter Cmax | 4 months
  Following completion of each cohort, bioanalytical and the PK parameter Cmax will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Eastenson, MD, Principal Investigator — Prism Research Clinic
Locations (1):
- Prism Clinical Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No